CLINICAL TRIAL: NCT02025023
Title: Local 5-Fluorouracil Injection for the Treatment of Chalazia: A Prospective, Comparative Study
Acronym: CTS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Matthew Zhang, Assistant Professor of Ophthalmology, University of Washington
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003748
Record Dates: First submitted 2013-12-29; First posted 2013-12-31 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Chalazion
Keywords: Size; Pain; Resolution; Complications; Swelling
MeSH Terms: conditions — Chalazion; Pain | interventions — Fluorouracil; Triamcinolone Acetonide; Triamcinolone; Curettage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Incision and Curettage (Active Comparator): A vertical incision over the area of chalazion will be done. Inflammatory material will be removed and the chalazion capsule will be excised.
  Interventions: Procedure: Incision and Curettage
- Injection of Triamcinolone Acetonide (Active Comparator): 0.1 ml of triamcinolone is injected directly in the chalazion.
  Interventions: Drug: Triamcinolone Acetonide; Procedure: Incision and Curettage
- Injection of 5-fluorouracil (Active Comparator): 0.1 ml of 5-fluorouracil is injected directly in the lesion transconjunctivally.
  Interventions: Drug: 5-fluorouracil Injection; Procedure: Incision and Curettage
- Injection of triamcinolone/5FU mixture (Active Comparator): 0.1 ml of a 4:1 mixture of 4 parts 5-FU and 1 part triamcinolone is injected in the lesion.
  Interventions: Procedure: Incision and Curettage; Drug: Triamcinolone Acetonide/5-fluorouracil mixture

INTERVENTIONS:
Drug: 5-fluorouracil Injection — If the chalazion is present at follow-up visit, another injection of 5-FU will be given.
  Other Names: 5-FU
  Arms: Injection of 5-fluorouracil
Drug: Triamcinolone Acetonide — If chalazion present at follow-up, another Triamcinolone injection will be done.
  Other Names: triamcinolone
  Arms: Injection of Triamcinolone Acetonide
Procedure: Incision and Curettage — If chalazion present at follow-up visit, patient will be randomized to receive local injection of either triamcinolone, 5-FU, or triamcinolone/5-FU mixture.
Drug: Triamcinolone Acetonide/5-fluorouracil mixture — If chalazion persists at follow-up visit, another injection of triamcinolone/5-FU mixture will be done.
  Arms: Injection of triamcinolone/5FU mixture

SUMMARY:
Local injection of 5-fluorouracil into a chalazion (stye) is as effective as local injection of triamcinolone (steroid) and incision and curettage for treatment of chalazia.

DETAILED DESCRIPTION:
This is a prospective randomized interventional study comparing four current standard-of-care treatments for chalazia: incision and curettage, local injection of triamcinolone, local injection of 5-FU, and local injection of combination triamcinolone/5-FU.

ELIGIBILITY:
Inclusion Criteria:

* Single or multiple chalazia in a single eyelid

Exclusion Criteria:

* Chalazia present for less than one month and no previous injection or incision and curettage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-12; Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Size of chalazion | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M Zhang, MD, Principal Investigator — University of Washington Eye Institute
Locations (1):
- University of Washington Eye Institute at Harborview, Seattle, Washington, United States